CLINICAL TRIAL: NCT01574885
Title: Double-blind, Randomized, Placebo Controlled Study Evaluating the Efficacy of Aerosal® in the Treatment of Sub-Obstructive Adenotonsillar Hypertrophy and Related Diseases
Brief Title: Efficacy of Aerosal® in the Treatment of Sub-Obstructive Adenotonsillar Hypertrophy and Related Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Tecno Sun SRL (Industry)
Collaborators: Centro Studi Gised (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEROSAL3
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea; adenotonsillar hypertrophy; salt; sodium chloride
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerosal (Experimental): This arm include all patients treated with Aerosal®
  Interventions: Device: Halotherapy
- Placebo (Placebo Comparator): This arm include all patients treated with placebo
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Halotherapy — The treatment consist of 10 session of micronized iodized salt (sodium chloride) inhalation in a chamber that reproduces the environmental characteristics of a natural salt cave. Each daily session last 30 minutes.
  Other Names: aerosal; salt; sodium chloride
  Arms: Aerosal
Device: Placebo — The treatment consist of 10 sessions in a chamber that emulates the environmental characteristics of a natural salt cave but with no salt emanation. Each daily session last 30 minutes.
  Other Names: comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Aerosal® compared to a placebo treatment in the prognosis of sub-obstructive adenotonsillar hypertrophy present for at least six months.

ELIGIBILITY:
Inclusion Criteria:

* Sub-Obstructive Adenotonsillar Hypertrophy lasting from at least six months and associated with sleep disordered breathing (respiratory pauses or sleep-apnea) and/or recurrent sero-mucus otitis
* Suspension for more than 3 months from the date of any immunosuppressive treatments (cyclosporin, systemic steroids)

Exclusion Criteria:

* Patients with acute bronchopulmonary disease, tuberculosis, severe hypertension, hyperthyroidism, cancer (chemotherapy), intoxication, heart failure, bronchial asthma.
* Iodine allergy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline of adenotonsillar hypertrophy degree equal to or greater than 25% | 2 weeks (10 sessions), 14 weeks

SECONDARY OUTCOMES:
Change from baseline of hypoacusis equal to or greater than 10 dB | 2 weeks (10 sessions), 14 weeks
  Change from baseline of hypoacusis equal to or greater than 10 dB, detected at the frequencies of the tone range (5, 10, 20, 40 KHz)
Any change from baseline of tympanometry curve | 2 weeks (10 sessions), 14 weeks
  Any change from baseline of tympanometry, defined as the passage from curve type B to curve type C/A or from curve type C to curve type A
Any change from baseline of adenotonsillar hypertrophy degree | 2 weeks (10 sessions), 14 weeks
Any change from baseline of basal SpO2% levels | 2 weeks (10 sessions), 14 weeks
  Any change from baseline of basal SpO2% mean levels as assessed by pulse-oximetry
Any change from baseline of apnea index | 2 weeks (10 sessions), 14 weeks
  Any change from baseline of apnea events in an hour (apnea index), as assessed by pulse-oximetry
Any change from baseline of sleep time percentage with SpO2<95% | 2 weeks (10 sessions), 14 weeks
  Any change from baseline of sleep time percentage with SpO2 levels under 95%, as assessed by pulse-oximetry
Any change from baseline of hypoacusis | 2 weeks (10 sessions), 14 weeks
  Any change from baseline of hypoacusis, detected at the frequencies of the tone range (5, 10, 20, 40 KHz)
Number of reported adverse events | 2 weeks (10 sessions), 14 weeks
  Number of reported adverse events (AEs) during treatment period or after the end of treatment, if suspected to be related with it

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Gelardi, MD, Principal Investigator — University General Hospital Consortium of Bari
Locations (1):
- University General Hospital Consortium, Bari, Italy

REFERENCES:
- [Derived] Gelardi M, Iannuzzi L, Greco Miani A, Cazzaniga S, Naldi L, De Luca C, Quaranta N. Double-blind placebo-controlled randomized clinical trial on the efficacy of Aerosal in the treatment of sub-obstructive adenotonsillar hypertrophy and related diseases. Int J Pediatr Otorhinolaryngol. 2013 Nov;77(11):1818-24. doi: 10.1016/j.ijporl.2013.08.013. Epub 2013 Aug 22. PMID 24041858